CLINICAL TRIAL: NCT04634916
Title: A Prospective, Multi-Center Clinical Study of the BD® WavelinQ™ EndoAVF System for the Creation of Arteriovenous (AV) Fistula in Patients Requiring Dialysis
Brief Title: Post-market Surveillance Study of the BD® WavelinQ™ EndoAVF System
Acronym: CONNECT-AV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-18-002
Record Dates: First submitted 2020-11-09; First posted 2020-11-18 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Kidney Disease, End-Stage; End-stage Renal Disease; Arteriovenous Fistula
Keywords: EndoAVF
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- EndoAVF (Experimental)
  Interventions: Device: EndoAVF Creation

INTERVENTIONS:
Device: EndoAVF Creation — Subjects will have an endoAVF created using the WavelinQ EndoAVF System

SUMMARY:
A prospective, single-arm, multi-center post-market surveillance study of the BD® WavelinQ™ EndoAVF System for the Creation of Arteriovenous (AV) Fistula in Patients Requiring Dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be either male or non-pregnant female ≥ 18 years of age with an expected lifespan sufficient to allow for completion of all study procedures.
2. Subject must voluntarily sign and date the Informed Consent Form (ICF) prior to collection of study data or performance of study procedures.
3. Subject must be willing to comply with the protocol requirements, including clinical follow-up.
4. Subjects who have established, non-reversible kidney failure, who are currently on dialysis at screening or are in immediate need (within 6 months of endoAVF creation) of dialysis.
5. Target treatment vein diameter(s) for endoAVF creation ≥ 2.0 mm as measured via Duplex Ultrasound (DUS) or Venography.
6. Target treatment artery diameter ≥ 2.0 mm as measured via Duplex Ultrasound (DUS) or Arteriogram.
7. Subject has adequate collateral circulation to the hand, in the opinion of the Investigator.
8. At least one superficial outflow vein diameter ≥ 2.5 mm and in communication with the target creation site via a proximal forearm perforating vein.

Exclusion Criteria:

1. The subject is in a hypercoagulable state.
2. The subject has known bleeding diathesis.
3. The subject has insufficient cardiac output to support a native fistula in the opinion of the Investigator.
4. Known history of active intravenous drug abuse.
5. "Planned" major surgical procedure within 6 months following index procedure or major surgery within 30 days prior to index procedure.
6. The subject has a known allergy or hypersensitivity to contrast media which cannot be adequately pre-medicated.
7. The subject has known adverse effects to sedation and/or anesthesia which cannot be adequately pre-medicated.
8. Evidence of active infection on the day of the index procedure (temperature of ≥ 38.0° Celsius and/ or WBC of ≥ 12,000 cells/ μL, if collected).
9. The subject has another medical condition, which, in the opinion of the Investigator, may cause him/her to be non-compliant with the protocol, confound the data interpretation, or is associated with a life expectancy insufficient to allow for the completion of study procedures and follow-up.
10. The subject is currently participating in an investigational drug or another device study that has not completed the study treatment or that clinically interferes with the study endpoints. Note: Studies requiring extended follow-up visits for products that were investigational, but have since become commercially available, are not considered investigational studies.
11. The subject has central venous stenosis or central vein narrowing > 50% based on imaging on the same side as the planned endoAVF creation.
12. Absence of a proximal forearm perforating vein feeding the target cannulation vein(s) from the target creation site via Duplex Ultrasound (DUS) or Venography.
13. Occlusion or stenosis > 50% of target cannulation vein(s) such as cephalic, median cubital, basilic, etc. assessed via Duplex Ultrasound (DUS) or Venography.
14. Significantly compromised venous or arterial flow in the treatment arm as determined by Investigator and Duplex Ultrasound (DUS) or Venography.
15. Presence of significant calcification at the target endoAVF location that could potentially impact the effectiveness of endoAVF creation as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Functional Cannulation Success | 6-months post index procedure
  The percentage of subjects dialyzed using successful 2-needle access of the endoAVF for at least 75% of dialysis sessions over a continuous 28-day period
Primary Patency | 6-months post index procedure
  Subjects maintaining primary patency of the endoAVF
Device- and procedure-related serious adverse events (SAE) | 30-days post index procedure
  Freedom from device-related or procedure-related SAEs

SECONDARY OUTCOMES:
Physiological Maturation | 2-weeks, 6-weeks, 6-months, and 24-months post index procedure
  Defined by duplex ultrasound flow in the brachial artery of at least 500ml/min and outflow vein diameter ≥ 4mm
Functional Maturation | 6-weeks, 3-, 6-, 12-, 18-, and 24-months post index procedure
  Successful prescribed dialysis with 2-needle cannulation of the endoAVF for three continuous weeks
Procedure Success | Index procedure
  Successful endoAVF creation
Cannulation Success | 6-weeks, 3-, 6-, 12-, 18-, and 24-months post index procedure
  Successful 2-needle endoAVF cannulation
Primary Patency | 6-weeks, 3-, 12-, 18-, and 24-months post index procedure
  Subjects maintaining primary patency of the endoAVF
Assisted Primary Patency | 6-weeks, 3-, 6-, 12-, 18-, and 24-months post index procedure
  Subjects maintaining assisted primary patency of the endoAVF
Secondary Patency | 6-weeks, 3-, 6-, 12-, 18-, and 24-months post index procedure
  Subjects maintaining secondary patency of the endoAVF
Functional Patency | through 24-months
  Interval of time from endoAVF cannulation success to involuntary access abandonment
Functional Cannulation Success | 3-, 12-, 18-, and 24-months post index procedure
  The percentage of subjects dialyzed using successful 2-needle access of the endoAVF for at least 75% of dialysis sessions over a continuous 28-day period
CVC Exposure/Use | 6-weeks, 3-, 6-, 12-, 18-, and 24-months post index procedure
Procedural Adjunctive Procedures | Index Procedure
  Adjunctive procedures performed at the time of the index procedure
Post Procedural Secondary Procedures | 2-weeks, 6-weeks, 3-, 6-, 12-, 18-, and 24-months post index procedure
  Number of secondary procedures conducted after the index procedure, broken down to identify interventions and second stage procedures

CONTACTS AND LOCATIONS:
Overall Officials: Eric Peden, MD, Principal Investigator — The Methodist Hospital Research Institute; Paul Kreienberg, MD, Principal Investigator — Albany Medical College
Locations (14):
- United States (14):
  - California Institute of Renal Research, La Jolla, California
  - San Francisco Vein & Vascular, San Francisco, California
  - Radiology and Imaging Specialists, Lakeland, Florida
  - Vascular and Interventional Specialists, Miami, Florida
  - UMass Chan School of Medicine, Worcester, Massachusetts
  - SSM St. Mary's, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - NC Nephrology, Raleigh, North Carolina
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Bluff City Vascular, Memphis, Tennessee
  - Baylor Scott & White, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No